CLINICAL TRIAL: NCT00617565
Title: A Multi-centre, Randomised, Parallel, Open Labelled Study to Compare the Efficacy and Safety Profile of Biphasic Insulin Aspart 30 (BIAsp 30) and Biphasic Human Insulin 30/70 (BHI 30/70) in Chinese Type 1 and 2 Diabetics
Brief Title: Efficacy and Safety of Biphasic Insulin Aspart 30 in Type 1 or 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1536
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
  Other Names: BIASP
Drug: biphasic human insulin

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate the efficacy of biphasic insulin aspart 30 on postprandial glycaemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes for at least 3 months
* Stabilised on current treatment with premixed human insulin for at least 4 weeks
* Body mass index (BMI) between 18-40 kg/m2
* HbA1c below 13.0%
* Able and willing to perform self-blood glucose monitoring

Exclusion Criteria:

* The receipt of any investigational drug within the last three months prior to this trial
* Has a history of drug abuse or alcohol dependence within the last 5 years
* Active proliferative retinopathy requiring laser or surgical intervention within the last year
* Recurrent major hypoglycaemia as judged by the Investigator
* Known or suspected allergy to trial product or related product

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2003-07-08 (Actual); Primary Completion 2003-11-26 (Actual); Study Completion 2003-11-26 (Actual)

PRIMARY OUTCOMES:
2-hr postprandial plasma glucose (PPPG) excursion | after 12 weeks of treatment

SECONDARY OUTCOMES:
HbA1c
Fasting plasma glucose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- China (3):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Beijing

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com